CLINICAL TRIAL: NCT00065702
Title: Biomarkers of Homeopathy in Fibromyalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000315-01 (NIH); BellI
Record Dates: First submitted 2003-07-31; First posted 2003-08-01 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; homeopathy; EEG; EKG; chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

INTERVENTIONS:
Drug: Active liquid remedy

SUMMARY:
The purpose of this study is to evaluate the efficacy of individualized classical homeopathy in treatment of persons with fibromyalgia and to determine the usefulness of electroencephalographic and electrocardiographic measures to serve as markers of differences between active and placebo treatment.

ELIGIBILITY:
Inclusion criteria:

* ACR diagnosis of fibromyalgia;
* Willing to take daily active or placebo liquid remedy under double blind conditions for 6 months, involving daily succussion and dilution of source liquid from a stock bottle;
* Willingness/ability to comply with dietary and lifestyle restrictions, i.e., no coffee in any form, no comphor or menthol-containing products; no electric blankets, no strong aromatics, no routine vaccinations, no concomitant use of acupuncture, chiropractic, polarity therapy, psychic healing, or magnet therapy;
* No dental drilling, MRI scans unless emergent;
* Withhold food or drink 30 mins before/after therapy;
* Stable conventional care for 2 months prior to entry;
* Willing to undergo 3 diagnostic physical exams, and to permit videotaping of interview sessions;
* Willing to fill out questionnaires

Exclusion criteria:

* Steroid-dependent medical conditions;
* Chronic benzodiazepine or anticonvulsant use;
* Use of tricyclic antidepressants, antihypertensives, and other drugs that alter orthostasis;
* Pregnancy;
* History of seizure disorder or syncope;
* Life-threatening medical conditions;
* Current active asthma;
* History of anaphylactic shock;
* Insulin-dependent diabetes;
* Active suicidal ideation or psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2000-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Iris R. Bell, MD, PhD, Principal Investigator — University of Arizona College of Medicine
Locations (1):
- U of Arizona College of Medicine, Program in Integrative Medicine, Tucson, Arizona, United States